CLINICAL TRIAL: NCT02160925
Title: Study of 99mTc-Sestamibi SPECT/CT Imaging for the Preoperative Diagnosis of Renal Oncocytoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00027784
Record Dates: First submitted 2014-06-06; First posted 2014-06-11 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Clinical T1 Renal Mass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preoperative 99mTc-Sestamibi SPECT/CT (Experimental)
  Interventions: Other: Preoperative 99mTc-Sestamibi SPECT/CT

INTERVENTIONS:
Other: Preoperative 99mTc-Sestamibi SPECT/CT

SUMMARY:
The objective of this study is to investigate the utility of 99mTc-sestamibi SPECT/CT imaging for the diagnosis of renal oncocytomas.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a solid enhancing cT1 renal mass detected on cross-sectional imaging
* Scheduled to undergo surgery with either partial or radical nephrectomy
* Age ≥18 years

Exclusion Criteria:

* Pregnancy
* Evidence of nodal or distant metastases
* History of other malignancy with concern for renal metastasis
* Known allergy to technetium or sestamibi

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2014-05; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Correlation of preoperative 99mTc-sestamibi SPECT/CT findings with tumor histology following surgical resection. | Within 2 weeks of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Allaf, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States